CLINICAL TRIAL: NCT04508439
Title: Effect of the Use of Anticoagulant Therapy During Hospitalization and Discharge in Patients With COVID-19 Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Regional de Alta especialidad de Ixtapaluca (Other)
Responsible Party: Principal Investigator, Omar Ramos-Peñafiel, Principal Investigator, Hospital Regional de Alta especialidad de Ixtapaluca
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NR-CEI-HRAEI-19-2020
Record Dates: First submitted 2020-08-05; First posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Covid19; Pneumonia; Coagulation Disorder; Pulmonary Embolism
Keywords: Covid-19; Mortality; anticoagulants; Deep venous thrombosis; Pulmonary embolism
MeSH Terms: conditions — COVID-19; Pneumonia; Hemostatic Disorders; Pulmonary Embolism; Venous Thrombosis | interventions — Enoxaparin; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Intervention Model Description: * Initially they will be randomized into two blocks, the first based on prophylactic Enoxaparin (Numbers 1 to 64) and the second (Numbers 65 to 128) will be assigned to the Enoxaparin therapeutic regimen arm at doses of 1mg / kg/dose twice up to date
  * During hospitalization, the clinical evolution will be evaluated according to the requirements of mechanical ventilation, the reduction in D-Dimer levels and the clinical outcome (discharge or death).
  * Those patients who are discharged will be Randomized in two following treatment arms
  * The allocation of patients in the outpatient stage will be carried out randomly 1: 1 to receive Rivaroxaban 10mg PO every 24hrs or only clinical follow-up.
  * Follow-up of adverse events will be carried out in the Hematology outpatient clinic with a first consultation 15 days after discharge and a second consultation 30 days after discharge. With dimer D, ferritin, protein C, blood count, ESR and on day 30 with CAT.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic enexaparin (Experimental): Enoxaparin dose of 1mg / kg / dose twice daily
  Interventions: Drug: Enoxaparin
- Therapeutic Enoxaparin (Active Comparator): Enoxaparin dose of 1mg / kg / dose daily
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Enoxaparin — Identify the benefit of different doses of low molecular weight heparin (enoxaparin) on the established clinical response due to lack of ventilatory support, length of hospital stay or death in patients requiring hospital care for COVID-19 infection.
  Other Names: low molecular weight heparin

SUMMARY:
Viral infections provoke the systemic inflammatory response and cause an imbalance between the procoagulant and anticoagulant homeostatic mechanisms. Multiple pathogenic mechanisms are involved, including endothelial dysfunction, increased von Willebrand factor, Toll receptor activation, and tissue factor pathway activation. D-dimer levels greater than 1000 ng / mL are associated with an 18-fold increased risk of mortality. In this context, many patients may require prophylaxis or antithrombotic treatment with low molecular weight heparins. Currently, there is no validated scheme on the dose and timing of the use of antithrombotic drugs.

The study aims to identify the effect of two anticoagulant strategies (prophylactic and therapeutic) on the progression to ventilatory support or death in patients with COVID-19 infection who require hospital care.

DETAILED DESCRIPTION:
Randomized clinical trial in patients with a confirmed infection by COVID-19 who require hospital treatment and subsequent ambulatory surveillance.

Study population. Patients with a diagnosis by PCR of COVID 19, over 18 years of age from the High Specialty Hospital of Ixtapaluca, who meet the inclusion criteria.

Statistic analysis. The student's T-test was carried out to identify the difference in the means of the quantitative variables between the groups. A value of P ≤ 0.05, 95% CI will be considered significant. For the hypothesis test, the chi-square test will be performed, considering a p≤ 0.05, 95% CI value to be significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of COVID-19 infection confirmed by polymerase chain reaction test (RQ-PCR) requiring hospital care for the administration of supplemental oxygen

Exclusion Criteria:

* Patients with life expectancy less than 48hrs
* Patients who require ventilatory support upon admission
* Age over 75 years or with a history of atrial fibrillation
* History of venous or arterial thrombosis
* Severe neurological impairment
* Absence of a primary caregiver to supervise the administration of medication
* History of cerebral hemorrhage
* History of previous use of oral anticoagulants
* History of major surgery 30 days prior to admission
* Uncontrolled systemic arterial hypertension
* KDIGO stage III chronic kidney disease or less
* Hemodialysis or peritoneal dialysis treatment
* History of active or inactive cancer
* Pregnant or postpartum patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-06-20 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
low molecular weight heparin (enoxaparin) and ventilatory support time | 30 days
  Identify the benefit of different doses of low molecular weight heparin (enoxaparin) on ventilatory support time in patients requiring hospital care for COVID-19 infection.
thrombotic complications and Rivaroxaban | 30 days
  To compare oral anticoagulation therapy by administering Rivaroxaban 10mg PO every 24 hours on early thrombotic complications
low molecular weight heparin (enoxaparin) and length of hospital stay | 30 days
  Identify the benefit of different doses of low molecular weight heparin (enoxaparin) on the length of hospital stay in patients requiring hospital care for COVID-19 infection.
low molecular weight heparin (enoxaparin) and mortality rate | 30 days
  Identify the benefit of different doses of low molecular weight heparin (enoxaparin) over mortality rate in patients requiring hospital care for COVID-19 infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Regional de Alta Especialidad de Ixtapaluca, Mexico City, Ixtapaluca, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Santos BC, Flumignan RL, Civile VT, Atallah AN, Nakano LC. Prophylactic anticoagulants for non-hospitalised people with COVID-19. Cochrane Database Syst Rev. 2023 Aug 16;8(8):CD015102. doi: 10.1002/14651858.CD015102.pub2. PMID 37591523